CLINICAL TRIAL: NCT01483547
Title: Reliability of Bispectral Index for Depth of Anesthesia Monitoring in Neurosurgical Patients
Brief Title: Reliability of BIS Monitoring in Neurosurgical Patients
Status: Completed | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Principal Investigator, Carla Carozzi, MD, Doctor, Dept. of Neuroanesthesia and Intensive Care, Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta
Other Study IDs: BISnch2011
Record Dates: First submitted 2011-11-25; First posted 2011-12-01 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Sovra and Intra Tentorial Lesions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Neurosurgical
  Interventions: Device: Bispectral Index (BIS Vista, Covidien)
- Non-neurosurgical
  Interventions: Device: Bispectral Index (BIS Vista, Covidien)

INTERVENTIONS:
Device: Bispectral Index (BIS Vista, Covidien) — BIS values at LOC, PI, ROC.

SUMMARY:
The aim of the study is to assess the reliability of Bispectral Index (BIS Vista , Covidien) in neurosurgical patients . BIS values at Loss of Consciousness (LOC), Post Intubation (PI) and Return of Consciousness (ROC) in neurosurgical patients are compared to those of non-neurosurgical patients, during routine anesthesia procedures.

ELIGIBILITY:
Inclusion Criteria:

* BIS > 90 at baseline (awake)
* ASA I or II

Exclusion Criteria:

* GSC < 15
* anticipated difficult ventilation and/or intubation
* BMI > 30
* surgical site that does not allow BIS monitoring
* bilateral hearing loss
* not speaking Italian Language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective craniotomy and elective spinal cord and column surgery.
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
BIS values at LOC, PI and ROC | 8 months

SECONDARY OUTCOMES:
incidence of intraoperative awareness | 0, 1, 3, 30 days after surgery
  intraoperative awareness assessed by BRICE Interview
incidence of postoperative delirium | 0, 1, 3, 30 days after surgery
  assessed by Nursing Delirium Scale and CAM-ICU.
predicted site effect drugs concentration at LOC, PI and ROC | 8 months
  Propofol and Remifentanil site effect concentrations delivered by TCI.
total amount of anesthetic drugs delivered at the end of surgery | 8 months
recovery time after surgery | 8 months
  Time needed for the patients to completely regain orientation

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Neurologico Carlo Besta, Milan, Milan, Italy